CLINICAL TRIAL: NCT00798590
Title: The Efficacy of GLP - 1 (7-36) Amide for Glycemic Control in Critically Ill Surgical Patients
Brief Title: The Efficacy of Glucagon Like Peptide (GLP) - 1(7-36) Amide for Glycemic Control in Critically Ill Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left JHU
Sponsor: Johns Hopkins University (Other)
Collaborators: Society of Critical Care Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00022551
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Critically Ill; Hypoglycemia
Keywords: Intensive insulin therapy (IIT); Insulin infusion; Tight glycemic control; Intensive Care Units
MeSH Terms: conditions — Critical Illness; Hypoglycemia | interventions — Glucagon-Like Peptide 1; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GLP-1 (Experimental)
  Interventions: Drug: Glucagon-Like Peptide-1
- Saline (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Glucagon-Like Peptide-1 — 5ng/kg-1/min-1 GLP-1 infused in 3 ml continuously over 72 hours.
  Other Names: GLP-1
  Arms: GLP-1
Drug: Saline — 5ng/kg-1/min-1 placebo infused in 3 ml continuously over 72 hours.
  Arms: Saline

SUMMARY:
The goal of this present proposal is to examine the efficacy of GLP-1 administered to control blood glucose in critically ill patients.

DETAILED DESCRIPTION:
All patients whom on admission to the ICU (surgical, burn, & cardiac) who are expected to receive intensive insulin therapy for at least 72 hours are eligible to be enrolled. Once enrolled, the patients will be randomized to one of two groups: the experimental (intravenous GLP-1 infusion for 72 hours) or control groups (intravenous 0.9% sodium chloride (NaCl) infusion for 72 hours) in a double masked fashion. While enrolled, all patients will receive standard-of-care insulin therapy. Both groups will be maintained on the standard ICU specific protocol for glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age > 21 to 75 years of age.
* All subjects who meet ICU specific criteria for inclusion in their glucose protocol and placed on insulin infusion protocol as standard of care.
* Able to obtain patient or proxy consent.

Exclusion Criteria:

* Current diagnosis of malignancy.
* Type 1 diabetes.
* Inability to obtain informed consent.
* On any Phase 1 trial.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-12; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dariush Elahi, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GLP-1 | Saline
Started | 11 | 8
Completed | 0 | 0
Not Completed | 11 | 8
Not completed — P.I, Left institution. Study terminated | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GLP-1 | Saline | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Customized [Number; unit: participants]
  >=21 and <=75 | 11 | 8 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 10 | 3 | 13
Region of Enrollment [Number; unit: participants]
  United States | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: To Compare the Composite Overall Amount of Insulin Used With GLP-1 vs. Placebo to Reach and Maintain the ICU-specific Target Glucose Range.
Time Frame: 2 years
Population: The PI left the institution and this study was terminated due to noncompliance with our Institutional Review Board. Outcome measure data, if collected, is unknown since no data are available.
Arm/Group | GLP-1 | Saline
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Compare the Number of Hypoglycemic Events Between GLP-1/Placebo Treatment
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | GLP-1 | Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The PI left the institution and this study was terminated due to noncompliance with our Institutional Review Board. Adverse event data, if collected, is unknown since no data are available.
Arm/Group | GLP-1 | Saline
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes